CLINICAL TRIAL: NCT00332098
Title: Family-Focused Treatment for Bipolar Adolescents
Brief Title: Effectiveness of Family-Focused Treatment Plus Pharmacotherapy for Bipolar Disorder in Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David J. Miklowitz, Ph.D., Professor of Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH073871 (NIH); R01MH073871 (NIH); R01MH073817 (NIH); R01MH074033 (NIH); DSIR 84-CTS (Registry Identifier: Division of Services and Intervention Research)
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Bipolar Disorder
Keywords: Childhood Mood Disorders; Family Treatment; Psychoeducation; Pharmacotherapy; Family Functioning; Psychosocial Intervention
MeSH Terms: conditions — Bipolar Disorder | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Family-Focused Treatment Plus Pharmacotherapy
  Interventions: Behavioral: Family-Focused Treatment Plus Pharmacotherapy
- 2 (Active Comparator): Enhanced Care Plus Pharmacotherapy
  Interventions: Behavioral: Enhanced Care Plus Pharmacotherapy

INTERVENTIONS:
Behavioral: Family-Focused Treatment Plus Pharmacotherapy — Participants assigned to FFT will take part in weekly treatment sessions with their families for 12 weeks, biweekly for 12 weeks, monthly for 3 months, and then trimonthly until Month 24. Medications used for the pharmacotherapy portion of the study will include mood stabilizers, such as lithium or divalproex sodium, and atypical antipsychotics, such as quetiapine. Participants will also receive anti-anxiety medications, psychostimulants, or antidepressants as needed.
  Arms: 1
Behavioral: Enhanced Care Plus Pharmacotherapy — Participants assigned to Enhanced Care will take part in weekly brief psychoeducation sessions for 3 weeks. The pharmacotherapy treatment will be the same as for the FFT participants.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of family-focused treatment (FFT) plus pharmacotherapy in treating adolescents with bipolar disorder.

DETAILED DESCRIPTION:
Bipolar disorder is a serious mental illness that causes drastic shifts in a person's mood, energy, and ability to function. Bipolar disorder can strike at any age, but it most commonly develops in late adolescence or early adulthood. The disorder is characterized by alternating episodes of mania and depression, often with periods of normal mood in between. Some symptoms of a manic episode include the following behaviors: increased energy, activity, and restlessness; excessively "high," overly good, euphoric mood; and extreme irritability. In contrast, a depressive episode is characterized by a lasting sad, anxious, or empty mood; feelings of hopelessness or pessimism; and decreased energy. Adolescents with bipolar disorder have high rates of disease recurrence, suicide attempts, functional impairment, and mental health service utilization, even with aggressive treatment with mood stabilizers and antipsychotic drugs. Research has suggested that FFT, a behavioral intervention consisting of psychoeducation, communication training, and problem solving training, may lead to improvements in mood symptoms in adolescents with bipolar disorder. This study will evaluate the effectiveness of FFT plus pharmacotherapy in treating adolescents with bipolar illness.

Participants in this 2-year, single-blind study will be randomly assigned to receive a combination of either FFT and pharmacotherapy or enhanced care and pharmacotherapy. Medications used for the pharmacotherapy portion of the study will include mood stabilizers, such as lithium or divalproex sodium, and atypical antipsychotics, such as quetiapine. Participants will also receive anti-anxiety medications, psychostimulants, or antidepressants as needed. All participants will receive pharmacotherapy for the full 2 years. Participants assigned to enhanced care will take part in weekly brief psychoeducation sessions for 3 weeks. Participants assigned to FFT will take part in weekly treatment sessions with their families for 12 weeks, biweekly for 12 weeks, monthly for 3 months, and then trimonthly until Month 24. Both FFT and enhanced care treatment sessions will include psychoeducation focusing on appropriate ways to manage bipolar disorder and its cycling nature. Crisis intervention sessions will also be offered to all participants on an as-needed basis for the duration of the study. Outcomes, including bipolar disorder symptoms, functioning, and service utilization, will be measured at study visits at Months 3, 6, 9, 12, 18, and 24.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 13 years, 0 months and 17 years, 11 months
* Meets The Diagnostic and Statistical Manual of Mental Disorders - IV criteria for either of the following conditions: bipolar I or bipolar II disorder with a manic, mixed, or hypomanic episode within 3 months of study entry; or a depressed episode within 3 months of study entry with a prior history of a manic, hypomanic, or mixed episode (if the participant only meets criteria for a current hypomanic episode, there must also be a history of at least one prior depressive, manic, or mixed episode)
* Has experienced severe depression, hypomania, or mania symptoms for a period of at least 1 week within the 3 months prior to study entry
* Lives with at least one biological or step-parent who is available and willing to participate in treatment (parents not currently living with the adolescent participant may also participate)

Exclusion Criteria:

* Currently in full recovery (experienced minimal symptoms for at least 8 continuous weeks)
* Meets Diagnostic and Statistical Manual of Mental Disorders, IV criteria for substance abuse disorder or substance dependence disorder within 3 months of study entry (based on the Kiddie Schedule for Affective Disorders and Schizophrenia - Present and Lifetime Version )
* Meets current criteria for bipolar, not otherwise specified, or substance-induced mood disorder
* Diagnosis of mental retardation, autism, or organic central nervous system disorder
* Severe, unremitting psychosis that is unresponsive to neuroleptic medications, and has lasted more than 3 months
* Requires extended inpatient treatment (although participant can be hospitalized at the time of intake into the study)
* Current life-threatening eating disorder, neurological condition, or other medical problem that requires immediate treatment
* Exhibits or expresses serious homicidal tendencies
* Victim of current sexual or physical abuse by parents or is in an environment marked by domestic violence among the parents or step-parents

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2006-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Time to recovery | Measured at Month 24
Time to recurrence | Measured at Month 24
Severity of manic and depressive symptoms | Measured at Month 24

SECONDARY OUTCOMES:
Functioning | Measured at Month 24
Quality of life | Measured at Month 24
Service utilization | Measured at Month 24

CONTACTS AND LOCATIONS:
Overall Officials: David J. Miklowitz, PhD, Principal Investigator — University of Colorado at Boulder; Robert A. Kowatch, MD, Principal Investigator — University of Cincinnati; David A. Axelson, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (3):
- United States (3):
  - University of Colorado, Dept. of Psychology, Boulder, Colorado
  - Cincinnati Children's Hospital Medical Center/MLC 3014, Cincinnati, Ohio
  - University of Pittsburgh Medical Center Western Psychiatric Institute, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Miklowitz DJ, George EL, Axelson DA, Kim EY, Birmaher B, Schneck C, Beresford C, Craighead WE, Brent DA. Family-focused treatment for adolescents with bipolar disorder. J Affect Disord. 2004 Oct;82 Suppl 1(Suppl 1):S113-28. doi: 10.1016/j.jad.2004.05.020. PMID 15571785
- [Background] Miklowitz DJ, Axelson DA, Birmaher B, George EL, Taylor DO, Schneck CD, Beresford CA, Dickinson LM, Craighead WE, Brent DA. Family-focused treatment for adolescents with bipolar disorder: results of a 2-year randomized trial. Arch Gen Psychiatry. 2008 Sep;65(9):1053-61. doi: 10.1001/archpsyc.65.9.1053. PMID 18762591
- [Result] Miklowitz DJ, Schneck CD, George EL, Taylor DO, Sugar CA, Birmaher B, Kowatch RA, DelBello MP, Axelson DA. Pharmacotherapy and family-focused treatment for adolescents with bipolar I and II disorders: a 2-year randomized trial. Am J Psychiatry. 2014 Jun;171(6):658-67. doi: 10.1176/appi.ajp.2014.13081130. PMID 24626789
- [Derived] O'Donnell LA, Weintraub MJ, Ellis AJ, Axelson DA, Kowatch RA, Schneck CD, Miklowitz DJ. A Randomized Comparison of Two Psychosocial Interventions on Family Functioning in Adolescents with Bipolar Disorder. Fam Process. 2020 Jun;59(2):376-389. doi: 10.1111/famp.12521. Epub 2020 Feb 3. PMID 32012257
- [Derived] Weintraub MJ, Schneck CD, Axelson DA, Birmaher B, Kowatch RA, Miklowitz DJ. Classifying Mood Symptom Trajectories in Adolescents With Bipolar Disorder. J Am Acad Child Adolesc Psychiatry. 2020 Mar;59(3):381-390. doi: 10.1016/j.jaac.2019.04.028. Epub 2019 May 28. PMID 31150753
- [Derived] O'Donnell LA, Axelson DA, Kowatch RA, Schneck CD, Sugar CA, Miklowitz DJ. Enhancing quality of life among adolescents with bipolar disorder: A randomized trial of two psychosocial interventions. J Affect Disord. 2017 Sep;219:201-208. doi: 10.1016/j.jad.2017.04.039. Epub 2017 Apr 28. PMID 28570966
- [Derived] Keenan-Miller D, Peris T, Axelson D, Kowatch RA, Miklowitz DJ. Family functioning, social impairment, and symptoms among adolescents with bipolar disorder. J Am Acad Child Adolesc Psychiatry. 2012 Oct;51(10):1085-94. doi: 10.1016/j.jaac.2012.08.005. Epub 2012 Aug 28. PMID 23021483
- See also: Robert Sutherland Center for the Evaluation and Treatment of Bipolar Disorder, University of Colorado, Boulder — http://rdsfoundation.org